CLINICAL TRIAL: NCT00797316
Title: An 8-week Randomized, Double-blind, Parallel-group, Multi-center, Forced-titration Study to Evaluate the Efficacy and Safety of Aliskiren Plus HCTZ Compared to Aliskiren Monotherapy in Metabolic Syndrome Patients With Stage 2 Hypertension
Brief Title: Aliskiren Plus HCTZ Compared to Aliskiren in Metabolic Syndrome Patients With Stage 2 Systolic Hypertension
Acronym: AIMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2410
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Hypertension; Metabolic Syndrome; aliskiren; hydrochlorothiazide; systolic blood pressure; diastolic blood pressure; stage 2
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren plus Hydrochlorothiazide (Experimental): Aliskiren (150 mg) plus Hydrochlorothiazide (12.5 mg) for one week. Subsequently up-titrated to Aliskiren (300 mg) plus Hydrochlorothiazide (25 mg). Medication was taken once daily in oral form.
  Interventions: Drug: Aliskiren; Drug: Hydrochlorothiazide
- Aliskiren (Active Comparator): Aliskiren (150 mg) for one week. Subsequently up-titrated to Aliskiren (300 mg). Medication was taken once daily in oral form.
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg or 300 mg taken once daily in oral form
Drug: Hydrochlorothiazide — Hydrochlorothiazide 12.5 mg or 25 mg taken once daily in oral form.
  Arms: Aliskiren plus Hydrochlorothiazide

SUMMARY:
The purpose of the study is to evaluate the blood pressure lowering effect and safety of aliskiren in combination with Hydrochlorothiazide (HCTZ) compared to aliskiren monotherapy when given to metabolic syndrome patients with stage 2 systolic hypertension (mean sitting systolic blood pressure [msSBP] ≥ 160 mm Hg and < 200 mm Hg).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and able to participate in the study, and who give written informed consent before any assessment is performed.
* Male or female outpatients ≥ 18 years old.
* Patients with stage 2 systolic hypertension. Patients must have a msSBP ≥160 mmHg and <200 mmHg at Study Visit 5 (randomization).
* Patients who have stage 2 systolic hypertension that meet at least 2 additional components of the metabolic syndrome as defined by the National *Cholesterol Education program (NCEP) criteria:

  * Abdominal obesity (waist circumference > than 102 cm for men and > 88 cm for women)
  * Current triglycerides ≥ 150 mg/dL or medical treatment for this condition.
  * Current HDL- Cholesterol <40 mg/dL in men and <50 mg/dL in women or medical treatment for this condition.
  * Fasting glucose >100 mg/dL and <126 mg/dL

Exclusion Criteria:

* Office blood pressure measured by cuff (msDBP ≥ 110 mmHg and or msSBP ≥ 200 mmHg) at any visit.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Use of aliskiren and/or a fixed dose combination of aliskiren HCTZ or participation in a clinical trial that had aliskiren and/or aliskiren HCTZ as treatment within 30 days of Visit 1.
* History of hypersensitivity to any of the medications or to drugs belonging to a similar therapeutic class (diuretics or renin inhibitors) as the study drugs.
* History or evidence of secondary form of hypertension.
* Refractory hypertension, defined as unresponsive to triple drug therapy at the maximum dose of each drug, one of which must be a diuretic, and not at blood pressure goal (140/90mmHg). Therapy with a fixed dose combination of two active substances represent two drugs.
* Patients on 4 or more antihypertensive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren/HCTZ: Aliskiren (150 mg) plus Hydrochlorothiazide (12.5 mg) for one week. Subsequently up-titrated to Aliskiren (300 mg) plus Hydrochlorothiazide (25 mg). Medication was taken once daily in oral form.
Period: Overall Study
Arm/Group | Aliskiren/HCTZ | Aliskiren
Started | 267 | 265
Completed | 244 | 233
Not Completed | 23 | 32
Not completed — Administrative problems | 1 | 0
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 4 | 8
Not completed — Protocol Deviation | 1 | 2
Not completed — Patient withdrew consent | 12 | 6
Not completed — Unsatisfactory therapeutic effect | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/HCTZ | Aliskiren | Total
Number analyzed (Participants) | 267 | 265 | 532
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.09) | 53.5 (10.87) | 53.9 (10.98)
Age, Customized [Number; unit: participants]
  < 65 | 217 | 233 | 450
  >= 65 | 50 | 32 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 129 | 257
  Male | 139 | 136 | 275

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Mean Sitting Systolic Blood Pressure (msSBP)
Time Frame: Baseline and Week 8
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/HCTZ | Aliskiren
Number analyzed (Participants) | 264 | 261
mm Hg | -30.38 (1.01) | -20.15 (1.01)

2. Secondary Outcome: Change From Baseline to Week 8 in Mean Sitting Diastolic Blood Pressure (msDBP)
Time Frame: 8 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/HCTZ | Aliskiren
Number analyzed (Participants) | 264 | 261
mm Hg | -11.26 (0.59) | -6.90 (0.60)

3. Secondary Outcome: Percentage of Participants With Blood Pressure Response at Week 8
Description: Response is defined as a patient with msSBP < 140 mmHg or a decrease from baseline ≥ 20 mmHg in msSBP during eight weeks of treatment.
Time Frame: 8 weeks
Population: full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren/HCTZ | Aliskiren
Number analyzed (Participants) | 264 | 261
Percentage of Participants | 78.4 | 55.2

4. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control at Week 8
Description: Blood pressure control is defined as a patient who achieves a target Blood Pressure of mean sitting Systolic Blood Pressure / mean sitting Diastolic Blood pressure < 140/90 mmHg.
Time Frame: 8 weeks
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren/HCTZ | Aliskiren
Number analyzed (Participants) | 264 | 261
Percentage of Participants | 58.7 | 34.5

5. Secondary Outcome: Change From Baseline to Week 8 in Pulse Pressure
Time Frame: Baseline and Week 8
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/HCTZ | Aliskiren
Number analyzed (Participants) | 264 | 261
mm Hg | -18.96 (0.74) | -13.33 (0.74)

ADVERSE EVENTS:
Arm/Group | Aliskiren/HCTZ | Aliskiren
Serious Adverse Events (participants affected / at risk) | 3/267 | 4/265
Other Adverse Events (participants affected / at risk) | 13/267 | 18/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/HCTZ (N=267) | Aliskiren (N=265)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/HCTZ (N=267) | Aliskiren (N=265)
Headache (Nervous system disorders) | 13 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.